CLINICAL TRIAL: NCT04908293
Title: A Comparison Between a Toothpaste With Micro Crystals of Hydroxyapatite and a Toothpaste With 1450 Ppm of Fluoride in the Home Remineralization of White Spot Lesions: a Clinical Trial.
Brief Title: Home Remineralization of White Spot Lesions With Two Different Toothpastes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-WHITESPOTS
Record Dates: First submitted 2021-05-23; First posted 2021-06-01 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: White Spot Lesion
Keywords: remineralization; hydroxyapatite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): Use of New Biorepair Advanced Sensitive toothpaste for home oral care.
  Interventions: Other: Biorepair toothpaste
- Control Group (Active Comparator): Use of Colgate toothpaste for home oral care.
  Interventions: Other: Colgate toothpaste

INTERVENTIONS:
Other: Biorepair toothpaste — Use of New Biorepair Advanced Sensitive for home oral care.
  Arms: Trial Group
Other: Colgate toothpaste — Use of Colgate toothpaste for home oral care.
  Arms: Control Group

SUMMARY:
The aim of the study is to compare white spot lesions before, during and after treatment with New Biorepair Advanced Sensitive toothpaste containing micro crystals of hydroxyapatite and Colgate toothpaste with 1450 ppm of fluoride. The timeline will consider the study begin, 15 days, 30 days and 90 days after the beginning of the study. The following indices will be recorded: BEWE Index, Schiff Air Index, VAS scale. After that, patients will fill in a satisfaction questionnaire.

DETAILED DESCRIPTION:
The aim of the study is to compare white spot lesions before, during and after treatment with two different toothpastes for home oral care. Patients who agree to sign the informed consent will be randomly assigned to two different groups:

* Trial Group will use New Biorepair Advanced Sensitive toothpaste containing micro crystals of hydroxyapatite;
* Control Group will use Colgate toothpaste with 1450 ppm of fluoride.

At the baseline, professional oral hygiene will be performed. The following indices will be recorded at the study begin and at the following 15, 30 and 90 days: BEWE Index, Schiff Air Index, VAS scale. After that, patients will fill in a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* patients with white spot lesions;
* patients with dental sensibility;
* adult patients;
* patients that sign the informed consent to participate to the study.

Exclusion Criteria:

* patients with low compliance or motivation to participate to the study;
* patients not presenting white spot lesions;
* patients with absence of dental sensibility;
* patients pregnant or breastfeeding;
* underage patients;
* patients with psychiatric diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Change of the BEWE Index - Basic Erosive Wear Examination (Barlet et al., 2008) | Study begin, 15, 30 and 90 days.
  Scoring criteria:
  0: no erosive tooth wear;
  1. initial loss of surface texture;
  2. distinct defect, hard tissue loss < 50% of the surface area;
  3. hard tissue loss ≥ 50% of the surface area.
Change in Schiff Air Index - Dental sensitivity test | Study begin, 15, 30 and 90 days.
  Scoring criteria:
  0: the subject did not respond to air blasting;
  1. the subject responded to air blasting;
  2. the subject responded to air blasting and requested discontinuation;
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change in VAS score | Study begin, 15, 30 and 90 days.
  Evaluation of the evoked pain with air blasting from 0 to 10. The VAS scale is a straight line with the endpoints defining extreme limits with "no pain at all"and "pain as bad as it could be"; they correspond respectively to 0 and 10. The patient indicates the score of the perceived pain from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.

REFERENCES:
- [Derived] Butera A, Gallo S, Pascadopoli M, Montasser MA, Abd El Latief MH, Modica GG, Scribante A. Home Oral Care with Biomimetic Hydroxyapatite vs. Conventional Fluoridated Toothpaste for the Remineralization and Desensitizing of White Spot Lesions: Randomized Clinical Trial. Int J Environ Res Public Health. 2022 Jul 16;19(14):8676. doi: 10.3390/ijerph19148676. PMID 35886524